CLINICAL TRIAL: NCT01500746
Title: Bedside Pulse Lavage Irrigation Project
Brief Title: Evaluation of the Effectiveness of Daily Pulse Lavage Therapy in Chronic Wounds
Acronym: PLI2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Robert Galiano, Assistant Professor of Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00057288
Record Dates: First submitted 2011-12-23; First posted 2011-12-28 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Wounds
Keywords: chronic wound treatment; pulse lavage; serial pulse lavage; wounds; bacterial colonization of wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lavage arm (Experimental): This group will serve as the experimental arm. They will undergo twice daily pulse lavage of their wounds for 4 days. In between the lavage treatments, their wounds will be dressed with moist gauze.
  Interventions: Procedure: Pulse lavage treatment
- Moist dressings (Active Comparator): This group will serve as the control group. They will undergo twice daily dressing changes with moist gauze dressings for a total of 4 days (8 dressing changes). Bacterial counts and gene expression analysis will be performed prior to the first dressing change and after the last dressing change.
  Interventions: Other: Dressing changes

INTERVENTIONS:
Procedure: Pulse lavage treatment — A pulse lavage machine will be used to irrigate the wound with a total of 4 liters of water, twice daily, for a total of 4 days (8 treatments).
  Other Names: Pulsed lavage (Stryker Pulsavac Plus); Wound containment apparatus
  Arms: Lavage arm
Other: Dressing changes — Wounds will be treated with moist gauze dressing changes twice daily for a total of 4 days (8 treatments).
  Arms: Moist dressings

SUMMARY:
This study evaluates the effectiveness of pulse lavage therapy in decreasing bacterial counts in chronic wounds.

DETAILED DESCRIPTION:
Pulse lavage irrigation is an effective method of cleaning both acute and chronic wounds. The major drawback to pulse irrigation is that it is extremely messy and can easily contaminate the patient's surroundings, putting other patients and the person operating the device at risk. In order to obtain the benefits of pulse lavage, we have created a device that will contain the water spray from the lavage and protect both the patient and their surroundings. Due to the fact that frequent (multiple times daily) pulse lavage therapy has not been possible previously, it is unknown how effectively serial pulse lavage irrigation reduces bacterial counts. This study evaluates the effectiveness of serial pulse lavage therapy in decreasing bacterial counts in chronic wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a chronic wound (as defined by the wound being present for >30 days) located on any part of their body
2. The wound must be smaller than 10cm in greatest diameter.
3. Patients must have an expected remaining hospital duration of 4 days
4. Patients must be willing and able to comply with all study procedures

Exclusion Criteria:

1. Patients must not have undergone any surgical excisions or debridements of the wound in the past 30 days
2. The wound may not undergo any surgical procedures or other treatments other than the study treatments during the course of the study.
3. The wound may not require any immediate surgical intervention or debridement
4. Patients may not start any new antibiotic therapy during the course of the study
5. Must not have an allergy to skin adhesives.
6. Patients must not be taking any immunosuppressive medications.
7. Subjects who, in the opinion of the investigator, may not complete the study for any reason.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Galiano, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Brown LL, Shelton HT, Bornside GH, Cohn I Jr. Evaluation of wound irrigation by pulsatile jet and conventional methods. Ann Surg. 1978 Feb;187(2):170-3. doi: 10.1097/00000658-197802000-00013. PMID 343735
- [Background] Granick MS, Tenenhaus M, Knox KR, Ulm JP. Comparison of wound irrigation and tangential hydrodissection in bacterial clearance of contaminated wounds: results of a randomized, controlled clinical study. Ostomy Wound Manage. 2007 Apr;53(4):64-6, 68-70, 72. PMID 17449917
- [Background] Kuehn BM. Chronic wound care guidelines issued. JAMA. 2007 Mar 7;297(9):938-9. doi: 10.1001/jama.297.9.938. No abstract available. PMID 17341696
- [Background] Svoboda SJ, Bice TG, Gooden HA, Brooks DE, Thomas DB, Wenke JC. Comparison of bulb syringe and pulsed lavage irrigation with use of a bioluminescent musculoskeletal wound model. J Bone Joint Surg Am. 2006 Oct;88(10):2167-74. doi: 10.2106/JBJS.E.00248. PMID 17015593
- [Background] Keblish DJ, DeMaio M. Early pulsatile lavage for the decontamination of combat wounds: historical review and point proposal. Mil Med. 1998 Dec;163(12):844-6. PMID 9866365
- [Background] Luedtke-Hoffmann KA, Schafer DS. Pulsed lavage in wound cleansing. Phys Ther. 2000 Mar;80(3):292-300. No abstract available. PMID 10696155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates extended from december 2011 to October 2013.
Period: Overall Study
Arm/Group | Lavage Arm | Moist Dressings
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lavage Arm | Moist Dressings | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants] — Northwestern Memorial Hospital, Chicago, IL
  participants
    United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Bacterial Counts
Description: A punch biopsy of the wound will be taken once the subject is enrolled in the study. A repeat biopsy will be taken after the 8th lavage treatment or the 8th dressing change. These will be sent for bacterial count analysis and the difference in bacterial counts will be evaluated. The lavage fluid from baseline measurements will be filtered and sent for bacterial counts and will be compared to the filtered fluid from the last lavage treatment. In addition, surface swabs will be taken at the beginning and end of the study and will be sent for bacterial counts as well. Bacterial counts from these lavage, biopsy specimen, and swabs will be averaged and analyzed.
Time Frame: Baseline and at 4 days
Measure: Mean (Full Range); unit: cfu/mL
Arm/Group | Lavage Arm | Moist Dressings
Number analyzed (Participants) | 4 | 4
cfu/mL | 4460 [-153 to 4580] | -1030000 [-1100000 to 158480]

2. Primary Outcome: Change in Gene Expression Analysis
Description: A punch biopsy will be taken at the beginning of the study. this will be sent for gene expression analysis. A repeat biopsy at the end of the study will also be sent at the end of the study, and a change in gene expression in analysis will be evaluated.
Time Frame: 4 days
Reporting Status: Not Posted

3. Secondary Outcome: Pain With Lavage Treatments
Description: After each lavage treatment, the subjects will complete a visual analogue scale that will determine the level of discomfort that they experienced during the study.
Time Frame: 4 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Lavage Arm | Moist Dressings
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No